CLINICAL TRIAL: NCT01378741
Title: Reducing Delirium After Cardiac Surgery: A Multifaceted Approach Of Perioperative Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: UHN10-0771A
Record Dates: First submitted 2011-06-20; First posted 2011-06-22 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Delirium; Cardiac Disease
Keywords: delirium; cardiac surgery; postoperative sedation
MeSH Terms: conditions — Delirium; Heart Diseases | interventions — Propofol; Dexmedetomidine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propofol (Active Comparator): Upon arrival to ICU patients will receive a propofol 2-6mg/kg infusion until tracheal extubation
  Interventions: Drug: Propofol
- Dexmedetomidine (Active Comparator): Upon arrival to ICU patients will receive dexmedetomidine bolus of 0.4mcg/kg followed by an infusion of 0.2-0.7mcg/kg per hour for a maximum period of 24 hours.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Propofol — Upon arrival to ICU patients will receive a propofol 2-6mg/kg infusion until tracheal extubation
  Other Names: Diprivan
  Arms: Propofol
Drug: Dexmedetomidine — Upon arrival to ICU patients will receive dexmedetomidine bolus of 0.4mcg/kg followed by an infusion of 0.2-0.7mcg/kg per hour for a maximum period of 24 hours.
  Other Names: Precedex
  Arms: Dexmedetomidine

SUMMARY:
The objective of this study is to reduce the incidence of postoperative delirium after cardiac surgery in the elderly patient. This proposal is a clinical trial designed to reduce delirium in patients undergoing cardiac surgery by replacing standard postoperative sedation protocols (propofol, midazolam, opioids) with a new alpha2-adrenergic receptor agonist (dexmedetomidine) possessing sedative, analgesic, and antinociceptive properties. Resource utilization analysis will be performed to determine cost effectiveness of the new treatment modality.

DETAILED DESCRIPTION:
The proposed study will be a prospective, randomized, open label study comparing multimodal protocols for postoperative sedation after cardiac surgery. Patients will be randomly allocated to either dexmedetomidine or propofol (control) groups according to a computer generated randomization code in predetermined size blocks of four.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥60 years, undergoing high risk cardiac surgery, signed informed consent.

Exclusion Criteria:

* Patients with symptomatic cerebrovascular disease, history of delirium, schizophrenia or preoperative use of psychotropic medications.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2011-04; Primary Completion 2014-07 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Dichotomous outcome, a number of patients with delirium in the two study groups. | up to 7 days postoperatively or discharge
  Assessment of delirium will be performed utilizing the CAM-ICU

SECONDARY OUTCOMES:
The total cost for each patient | Up to 7 days or discharge
  Summation of direct-variable, direct-fixed, and overhead costs

CONTACTS AND LOCATIONS:
Overall Officials: George Djaiani, MD, Principal Investigator — Toronto General Hospital, UHN
Locations (1):
- University Health Network, Toronto, Ontario, Canada